CLINICAL TRIAL: NCT03845894
Title: Single Injection Interscalene Brachial Plexus Nerve Block With Adjuvants vs. Liposomal Bupivacaine Interscalene Brachial Plexus Nerve Block for Total Shoulder Arthroplasty
Brief Title: Interscalene Block With Liposomal Bupivacaine vs. Interscalene Block With Bupivacaine and Adjuvants
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: feasibility
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00055981
Record Dates: First submitted 2019-01-22; First posted 2019-02-19 (Actual); Results first posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2022-09

CONDITIONS: Shoulder Arthroplasty
Keywords: Shoulder Replacement Surgery; Interscalene Nerve Block; Liposomal Bupivacaine; Shoulder pain; Regional anesthesia; Brachial plexus blockade
MeSH Terms: conditions — Shoulder Pain | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Liposomal Bupivacaine Interscalene brachial plexus (ISB) (Active Comparator)
  Interventions: Drug: Liposomal bupivacaine
- Bupivacaine with adjuvants ISB (Active Comparator)
  Interventions: Drug: Bupivacaine with adjuvants

INTERVENTIONS:
Drug: Liposomal bupivacaine — Interscalene brachial plexus blockade using liposomal bupivacaine (expanded with plain bupivacaine)
  Arms: Liposomal Bupivacaine Interscalene brachial plexus (ISB)
Drug: Bupivacaine with adjuvants — Interscalene brachial plexus blockade using plain bupivacaine with adjuvants: clonidine, epinephrine, buprenorphine, dexamethasone.
  Arms: Bupivacaine with adjuvants ISB

SUMMARY:
The purpose of this study is to determine whether the use of plain bupivacaine with common adjuvants for interscalene block (ISB) provides non-inferior analgesic results compared to the use of liposomal bupivacaine for ISB, in patients undergoing total shoulder arthroplasty.

DETAILED DESCRIPTION:
The primary objective of this clinical study is to evaluate the comparative efficacy of interscalene block (ISB) using plain bupivacaine with adjuvants vs. liposomal bupivacaine on mean postoperative pain levels in patients who have undergone a total shoulder arthroplasty within the first 48 hours. Principal Investigators hypothesize that ISB using plain bupivacaine with adjuvants will provide similar pain relief as ISB using liposomal bupivacaine.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing total shoulder arthroplasty (not a reverse)
* Age ≥ 18 years
* Ability to understand and the willingness to sign an IRB-approved informed consent document.
* ASA patient status I-III patients
* Weight Greater than or equal to 50 kg

Exclusion Criteria:

* Contraindications to an interscalene block or phrenic blockade
* Infection at injection site
* Pre-existing neurological dysfunction affecting the operative extremity
* Chronic pain diagnosis or opioid use >40mg oxycodone daily equivalents or use of long-acting opioids
* BMI >40
* Uncontrolled diabetes (A1c >8.0)
* Concurrent painful physical condition requiring analgesic treatment (eg, NSAID or opioid) in the postsurgical period for pain not strictly related to the surgery
* Contraindications to any pain-control agents planned for surgical or postsurgical use (i.e., bupivacaine, hydromorphone, etc.)
* Patients who are wards of the state
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to bupivacaine or liposomal bupivacaine.
* Patients with moderate-severe hepatic or renal impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2022-06-25 (Actual); Study Completion 2022-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doug Jaffe, DO, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Will be shared upon request: raw data and statistical calculations
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Available after study conclusion, for up to 3 years afterward.

REFERENCES:
- [Background] Sakamoto B, Keiser S, Meldrum R, Harker G, Freese A. Efficacy of Liposomal Bupivacaine Infiltration on the Management of Total Knee Arthroplasty. JAMA Surg. 2017 Jan 1;152(1):90-95. doi: 10.1001/jamasurg.2016.3474. PMID 27732710
- [Background] Hamilton TW, Athanassoglou V, Mellon S, Strickland LH, Trivella M, Murray D, Pandit HG. Liposomal bupivacaine infiltration at the surgical site for the management of postoperative pain. Cochrane Database Syst Rev. 2017 Feb 1;2(2):CD011419. doi: 10.1002/14651858.CD011419.pub2. PMID 28146271
- [Background] Pichler L, Poeran J, Zubizarreta N, Cozowicz C, Sun EC, Mazumdar M, Memtsoudis SG. Liposomal Bupivacaine Does Not Reduce Inpatient Opioid Prescription or Related Complications after Knee Arthroplasty: A Database Analysis. Anesthesiology. 2018 Oct;129(4):689-699. doi: 10.1097/ALN.0000000000002267. PMID 29787389
- [Background] Hamilton TW, Athanassoglou V, Trivella M, Strickland LH, Mellon S, Murray D, Pandit HG. Liposomal bupivacaine peripheral nerve block for the management of postoperative pain. Cochrane Database Syst Rev. 2016 Aug 25;2016(8):CD011476. doi: 10.1002/14651858.CD011476.pub2. PMID 27558150
- [Background] Rabin T. FDA In Brief: FDA approves new use of Exparel for nerve block pain relief following shoulder surgeries.

RESULTS

PARTICIPANT FLOW:
Groups:
- Liposomal Bupivacaine ISB: Liposomal bupivacaine: Interscalene brachial plexus blockade using liposomal bupivacaine (expanded with plain bupivacaine)
Period: Overall Study
Arm/Group | Liposomal Bupivacaine ISB | Bupivacaine With Adjuvants ISB
Started | 12 | 13
Completed | 12 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liposomal Bupivacaine ISB | Bupivacaine With Adjuvants ISB | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 6 | 8
  >=65 years | 10 | 7 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 8 | 7 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 12 | 11 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 10 | 9 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 12 | 13 | 25

OUTCOME MEASURES:

1. Primary Outcome: Average Pain Scores for the First 48 Hours
Description: Pain levels will be measured by the mean Visual Analogue Scale- Numeric Rating Scale (VAS-NRS). The VAS-NRS is an 11 point scale with 0 (no pain) to 10 (worst possible pain). Higher scores denote worse outcome.
Time Frame: At 48 hours postoperatively
Population: The software interface in this website will not allow for AUC as an acceptable outcome to satisfy field entries. Therefore, here the AUC is not reported here, but rather then mean and standard deviation are reported.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Liposomal Bupivacaine ISB | Bupivacaine With Adjuvants ISB
Number analyzed (Participants) | 12 | 13
units on a scale | 3.2 (2.0) | 3.6 (2.4)
Statistical Analysis 1: Comparison: Liposomal Bupivacaine ISB vs Bupivacaine With Adjuvants ISB; Test type: Non-Inferiority — There have been no studies to evaluate pain scores ISB w/ plain bupi+adjuvants. Power to detect difference at least 0.4 on the VAS scale. Threshold for inferiority is difference >=2 points on the VAS scale. Will use two-sample t test with α= 0.05 and β= 0.1. Postop opioid consumption, total post-op opioid @ 1st 48 hours in oxycodone equivalents. Mean opioid consumption per cohort is calculated, & the cohorts compared for statistical difference with two-sample t test, with α= 0.05 and β= 0.1; p = 0.14, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Postoperative Opioid Consumption for the First 48 Hours
Description: Morphine milligram equivalents (MME) over a 48 hour period
Time Frame: up to 48 hours
Measure: Mean (Standard Deviation); unit: Morphine milligram equivalents (MME)
Arm/Group | Liposomal Bupivacaine ISB | Bupivacaine With Adjuvants ISB
Number analyzed (Participants) | 12 | 13
Morphine milligram equivalents (MME) | 22.9 (20.6) | 28.5 (23)

3. Secondary Outcome: Satisfaction With Surgical Experience
Description: Satisfaction scale is from 1-5, with the higher score being highest level of satisfaction
Time Frame: at 48 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Liposomal Bupivacaine ISB | Bupivacaine With Adjuvants ISB
Number analyzed (Participants) | 12 | 13
units on a scale | 4.75 (.45) | 3.46 (1.56)

ADVERSE EVENTS:
Time Frame: 24 hours
Description: events that occurred during first 24 hours after surgery
Arm/Group | Liposomal Bupivacaine ISB | Bupivacaine With Adjuvants ISB
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13
Other Adverse Events (participants affected / at risk) | 0/12 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/94/NCT03845894/Prot_SAP_001.pdf
  • Informed Consent Form (2022-04-05): https://cdn.clinicaltrials.gov/large-docs/94/NCT03845894/ICF_000.pdf